CLINICAL TRIAL: NCT03525314
Title: Development of Achilles Tendon Elongation and Its Effect on Physical Function the First Year After Rupture: A Prospective Cohort Study
Brief Title: Development of Achilles Tendon Elongation and Its Effect on Physical Function the First Year After Rupture
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Maria Swennergren Hansen, Principal Investigator, Hvidovre University Hospital
Other Study IDs: Achilles HVH Cohort
Record Dates: First submitted 2018-05-03; First posted 2018-05-15 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to examine how elongation of the Achilles tendon develops during the first year after rupture among patients with an Achilles tendon rupture, and how it affects physical function.

The aim is to define a cutoff of acceptable elongation dividing the patients who obtain normal physical function (Limb Symmetry Index > 90%) from those who do not.

Patients treated both operatively and non-operatively will be included.

ELIGIBILITY:
Inclusion Criteria:

* Appointment in the Outpatients Department within 4 days of injury.
* Total Achilles tendon rupture.
* Initial treatment with split cast with the ankle in maximal plantar flexion must be started within 24 hours of injury.
* The patient must be expected to be able to attend rehabilitation and postexaminations.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.

Exclusion Criteria:

* Rupture of the Achilles tendon either at the insertion on the calcaneus or at musculotendinous junction of the triceps surae.
* Previous rupture of the Achilles tendon in any of the two legs.
* Treated with Fluorquinolons or corticosteroids within the last 6 months.
* In medical treatment of diabetes.
* Suffers from rheumatic disease.
* Other conditions prior to the injury resulting in reduced function of any of the two legs.
* Contra-indication for surgery: severe arthrosclerosis with no palpable pulse in the foot, broken skin in the Achilles region of the injured leg.
* Inability to lie in prone position on the operating table.
* Terminal illness or severe medical illness: ASA (American Society of Anesthesiologists) score higher than or equal to 3.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients treated for acute Achilles tendon rupture at Amager-Hvidovre Hospital during the study period will be offered to participate in the study. The study cohort of study with uniqe clinical trials ID: Achilles HVH RCT is also included in this cohort.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Copenhagen Achilles Length Measure | Evaluation method after 12 months of started treatment
  The examination of both the total and the free part of the achilles tendon of both the injured and un-injured leg is performed. The free part of the achilles tendon is defined as the distance between the proximal border of calcaneus and the musculotendinous junction of the soleus muscle. The total length of the achilles tendon is the distance between the proximal border of calcaneus and the musculotendinous junction of the medial gastrocnemius muscle. Measurement is perfomed as described by Barfod et al (1).

SECONDARY OUTCOMES:
Copenhagen Achilles Length Measure | Evaluation method after 0-4 days, 3 weeks, 9 weeks, 4 months, 6 months of started treatment
  The examination of both the total and the free part of the achilles tendon of both the injured and un-injured leg is performed (the free part is measured from week 9). The free part of the achilles tendon is defined as the distance between the proximal border of calcaneus and the musculotendinous junction of the soleus muscle. The total length of the achilles tendon is the distance between the proximal border of calcaneus and the musculotendinous junction of the medial gastrocnemius muscle. Measurement is perfomed as described by Barfod et al (1).
Indirectly, clinical Achilles tendon length estimate | Evaluation method after 9 weeks, 4, 6 and 12 months of started treatment.
  Achilles tendon length is indirectly estimated clinically by use of the Achilles Tendon Resting Angle (ATRA) or the Achilles Tendon Length Measure (ATLM). The patient lies flat in prone position on the examination bed. The knee is flexed at 90 degrees and the ankle sits in relaxed position. The ATRA is determined as the angle between the corpus of the fibula and the corpus of the 5th metatarsus. The ATLM is determined as the distance from the caput of the 5th metatarsus to the surface of the examination bed. Both the ATRA and the ATLM are determined for both the injured and the uninjured leg. The difference between the healthy and the injured leg is evaluated.
Achilles tendon Total Rupture Score (ATRS) | Evaluation method after 0-4 days, 3 weeks, 9 weeks, 4, 6 and 12 months of started treatment
  Patients will fill out the ATRS questionnaire in connection to the follow-up visits in the Outpatients Department. ATRS is a patient-reported outcome measure.
  This questionnaire is a part of the usual examination of the patients' function, and is used during all follow-ups in the usual care.
Heel-rise Work test | Evaluation method after 4, 6 and 12 months of started treatment.
  An endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel rises are counted and measured and plotted into a diagram on an X-axis and Y-axis respectively. The results are then compared to the weight of the patient and the total work is estimated as area under the curve. The heel lift distance between the heel and the floor is measured in millimeters. The procedure is performed on the uninjured leg first and subsequently on the injured leg. The patient is barefoot for the heel-rise work test and stands on a flat surface with a 10 degree inclination. For these functional tests a measurement system MuscleLab (Ergotest Technology, Oslo, Norway) will be used.
Calf circumference | Evaluation method after 9 weeks, 4, 6 and 12 months of started treatment
  The patient is sits on an examination bed with legs hanging down. The circumference of the calf is measured using a measuring tape (13 cm under apex patella).
MRI | After 1 year of the started treatment
  MRI will be conducted to obtain a deeper understanding of how the different structures in the muscle-tendon complex change the first year after rupture. The MRI will be conducted at Copenhagen University Hospital Amager-Hvidovre in an Acanto 1,5 T scanner. Both lower legs will be scanned. The patient's head and upper-body are outside the scanner. Total time for the patient in the scanner is approximately 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Maria S Hansen, PT, MSc, Principal Investigator — Copenhagen University Hospital, Amager-Hvidovre
Locations (1):
- Department of Physiotherapy and Orthopedical surgery, Copenhagen University Hospital, Amager-Hvidovre, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
There is no plan of sharing data with researchers not already included in this study.

REFERENCES:
- [Background] Barfod KW, Riecke AF, Boesen A, Hansen P, Maier JF, Dossing S, Troelsen A. Validation of a novel ultrasound measurement of achilles tendon length. Knee Surg Sports Traumatol Arthrosc. 2015 Nov;23(11):3398-406. doi: 10.1007/s00167-014-3175-2. Epub 2014 Jul 20. PMID 25038882